CLINICAL TRIAL: NCT03721705
Title: A Randomized Pivotal Study of RenewTM NCP-5 for the Treatment of Mild Cognitive Impairment Due to Alzheimer's Disease or Mild Dementia of the Alzheimer's Type
Brief Title: Renew NCP-5 for the Treatment of Mild Cognitive Impairment Due to Alzheimer's Disease (AD) or Mild Dementia of the Alzheimer's Type
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Renew Research, LLC (Other)
Collaborators: Navitas Clinical Research, Inc (Unknown); ClinEdge (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RenewTM NCP-5-1001
Record Dates: First submitted 2018-08-01; First posted 2018-10-26 (Actual); Results first posted 2022-04-19 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-04

CONDITIONS: Alzheimer Disease; Cognitive Dysfunction; Mild Cognitive Impairment; Mild Dementia; Cognitive Decline; Dementia, Alzheimer Type
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to either the treatment group or the sham group.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Treatment Arm (Experimental): The first four sessions will be the escalation phase using the Renew NCP-5. There will be a 5-minute ramp up period where the pressure is increased 1 psi/min until the desired pressure is reached. The goal for the treatment group will be at least 2.5 psi for the first treatment, and then escalate the pressure gradually through the fourth session with an average goal of 3 psi/session. After the fourth session, the pressure will be slowly increased to reach the maximum level the subject can tolerate with a goal of reaching 3-6 psi.
  Interventions: Device: Renew NCP-5
- Sham Arm (Sham Comparator): The subjects will receive the same initial and maintenance treatment regimen on the Renew NCP-5. The pressure will not exceed an average of 0.5 psi over all treatments.
  Interventions: Device: Renew NCP-5

INTERVENTIONS:
Device: Renew NCP-5 — Treatment will be given 3-5 times a week for a total of 35 treatments over 12 weeks.

SUMMARY:
A Randomized Pivotal Study of RenewTM NCP-5 for the Treatment of Mild Cognitive Impairment due to Alzheimer's Disease or Mild Dementia of the Alzheimer's Type is a pivotal, single blind, parallel design, multi-site study intends to examine the efficacy and safety of RenewTM NCP-5 therapy in the treatment of Cognitive Impairment due to Alzheimer's Disease or Mild Dementia of the Alzheimer's Type. Subjects will be prospectively randomized to treatment or sham (in a 1:1 ratio) using stratification for Cognitive Impairment due to Alzheimer's Disease or Mild Dementia of the Alzheimer's Type, and Cardiovascular Risk (CVR) score at multiple sites. Subjects, ages 55-85, will be consented for 13 months and will receive thirty-five 60-minute RenewTM NCP-5 treatment sessions during a 7-to-12-week initial treatment period, and then transition to a lower frequency maintenance period (twice a week) for a total treatment period of 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Be 55-85 years of age at the time of signing the informed consent
2. Be able to provide consent or have legally authorized representative/caregiver who can provide consent
3. Be able to read and write in English or Spanish
4. Have a clinical diagnosis consistent with 2011 National Institute of Aging - Alzheimer's Association (NIA-AA) "core clinical criteria" guidelines for: (i) The diagnosis of dementia due to Alzheimer's disease or (ii) The diagnosis of mild cognitive impairment due to Alzheimer's disease:

   * Montreal Cognitive Assessment (MOCA) score of greater than or equal to 11
   * All required checkboxes within the study checklist for "The diagnosis of probable AD dementia" must be "yes" or
   * All required checkboxes within the study checklist for "The diagnosis of mild cognitive impairment due to Alzheimer's disease" must be "yes"
5. Stable medications for past 30 days and plan to remain on stable medications for the first 24 weeks of study participation for treatment of chronic conditions.
6. Subject should have a caregiver, study partner or companion (which can be a domestic party) and may conduct the assessment over the phone if they don't accompany the participant).
7. Must have the potential to improve by at least 2 points or more in the Vascular Dementia Assessment Scale cognitive subscale (vADAS-COG)

Exclusion Criteria:

1. Unwilling or unable to participate in study procedures
2. Weight >297 lbs. or >135 kg at screening
3. Major confounding neurodegenerative or psychiatric disorder unrelated to the condition under study, including:

   1. History of clinically-evident stroke
   2. Current uncontrolled epileptic seizures or epilepsy
   3. Multiple Sclerosis or Parkinson's Disease
   4. Current clinically significant major psychiatric disorder (e.g., Major Depressive Disorder) according to the Fifth Edition of Diagnostic and Statistical Manual of Mental Disorders (DSM-V) criteria or significant psychiatric symptoms (e.g., hallucinations) that could impair the completion of the study
4. Anyone with active or history of cerebral hemorrhage including subdural & subarachnoid or cerebral aneurysm
5. Evidence of any of the following (based on Section 4.1.1(D) of the 2011 NIA-AA guidelines on The diagnosis of dementia due to Alzheimer's disease):

   1. Substantial concomitant cerebrovascular disease, defined by a history of a stroke temporally related to the onset or worsening of cognitive impairment; or the presence of multiple or extensive infarcts or severe white matter hyperintensity burden
   2. Core features of Dementia with Lewy bodies other than dementia itself
   3. Prominent features of behavioral variant frontotemporal dementia
   4. Prominent features of semantic variant primary progressive aphasia or nonfluent/agrammatic variant primary progressive aphasia
   5. Evidence for another concurrent, active neurological disease, non-neurological medical comorbidity or use of medication that could have a substantial effect on cognition
6. In the opinion of the investigator, any current clinically-significant systemic illness or medical condition that is likely to result in deterioration of the subject's condition, affect the subject's safety during the study, or to be incompatible with performance of the study procedures, including:

   1. History of head trauma with a diagnosis of moderate to severe traumatic brain injury
   2. Known current substantially elevated intracranial pressure
   3. Known current significant sleep deprivation
   4. Known history (within five years) or current significant drug abuse or alcoholism
7. Any contraindication for MRI such as insulin pumps or pacemakers, including dual chamber pacemakers where atrial pacing may interfere with RenewTM NCP-5 inflation timing sequence
8. Hypotension as defined as <80/50 blood pressure at the time of screening
9. Ongoing uncontrolled severe hypertension (≥ 180 mmHg systolic or ≥ 110 mmHg diastolic
10. Heart rates < 35 or >125 beats per minute (BPM) at screening
11. Current uncontrolled arrhythmia. Controlled arrhythmia should have beat-to-beat, cycle-length variability less than ±25% at rest.
12. Current congestive heart failure
13. Cardiac catheterization within two weeks, any surgical intervention within six weeks before RenewTM NCP-5 treatment or a hip or knee replacement within 3 months as long as rehab is complete and symptoms have resolved.
14. Known presence of abdominal aortic aneurysm
15. Existing aortic insufficiency grade II or higher (regurgitation can prevent diastolic augmentation)
16. Current or past venous thrombosis or thromboembolism
17. Current limiting peripheral vascular disease with history strongly suggestive of lower extremity ischemia or claudication, arterial occlusive disease (aortoiliac, ileofemoral, or femoral popliteal)
18. Demonstrable deficiency in sensation in lower extremities as a result of diabetes or other medical condition
19. Current bleeding disorders.
20. Current use of major anti-coagulation therapy (such as Heparin therapy or Coumadin® therapy) with International Normalized Ratio (INR) > 1.5
21. Current severe pulmonary disease that prevents the subject from lying supine
22. Presence of local infection, vasculitis, burn, open wound, or bone fracture on any limb which would prevent the ability to perform the RenewTM NCP-5 treatment
23. Current use of medications that in the investigator's judgement are incompatible with the study goals
24. Significant changes in existing medical plans for treatment of cognitive impairment or dementia in last three months and/or or planned changes during the trial
25. Presence of any of the contraindications for using the RenewTM NCP-5 device
26. Athletic injuries, including Charley horses, pulled muscles and/or edematous muscles; necrotizing cellulitis in the past 30 days which would prevent the ability to perform the RenewTM NCP-5 treatment (evaluate and treat prior to RenewTM NCP-5 treatment)
27. Unwilling or unable to maintain stable exercise regimen throughout the trial
28. Participation in any clinical drug trial 30 days or five half-lives, whichever is longer, prior to screening visit
29. Use of any device to increase cerebral blood flow in the past 30 days.
30. History of claustrophobia.
31. Subject unable to lay supine for 90 minutes

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2018-11-12 (Actual); Primary Completion 2021-03-23 (Actual); Study Completion 2021-03-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Billy Tally, Study Director — Stage 2 Innovations
Locations (12):
- United States (10):
  - Xenoscience, Phoenix, Arizona
  - Irvine Clinical Research, Irvine, California
  - Charter Research, Lady Lake, Florida
  - Miami Dade Medical Research Institute, Miami, Florida
  - iResearch Atlanta, Atlanta, Georgia
  - iResearch Savannah, Savannah, Georgia
  - University of Kansas Medical Center, Kansas City, Kansas
  - Cardiovascular Advantages, LLC, Baton Rouge, Louisiana
  - Neuro-Behavioral Clinical Research, Canton, Ohio
  - Northwest Clinical Research Center, Bellevue, Washington
- St. James's Hospital, Dublin, Ireland
- National University Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment Arm | Sham Arm
Started | 95 | 95
Completed | 85 | 77
Not Completed | 10 | 18
Not completed — Adverse Event | 2 | 0
Not completed — Withdrawal by Subject | 4 | 10
Not completed — No Suitable Study Partner | 1 | 0
Not completed — Early Termination Due to Coronavirus Disease 2019 (COVID-19) | 3 | 7
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Arm | Sham Arm | Total
Number analyzed (Participants) | 95 | 95 | 190
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.5 (7.69) | 68.1 (7.20) | 68.3 (7.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 61 | 117
  Male | 39 | 34 | 73
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 17 | 35
  Not Hispanic or Latino | 77 | 78 | 155
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 3 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 13 | 13 | 26
  White | 76 | 78 | 154
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 95 | 93 | 188
  Ireland | 0 | 2 | 2
Mild Cognitive Impairment (MCI) due to AD [Count of Participants; unit: Participants] | 69 | 68 | 137
Mild AD [Count of Participants; unit: Participants] | 26 | 27 | 53
Low/Medium Cardiovascular Risk [Count of Participants; unit: Participants] | 62 | 61 | 123
High/Very High Cardiovascular Risk [Count of Participants; unit: Participants] | 33 | 34 | 67

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline to 24 Weeks in Vascular Dementia Assessment Scale Cognitive Subscale (vADAS-cog) Using the Average of Scores at 12, 18 and 24 Weeks.
Description: The vADAS-cog assessment includes 17 subscale scores. The total score is the sum of all scaled scored from 0-120. The higher values represent more cognitive impairment. The change in vADAS-cog scores from baseline at the timepoints of 12, 18, and 24 weeks is averaged together for each patient. The primary outcome measure is the average of those values for all patients in a group.
Time Frame: 24 weeks
Population: There were 7 treatment and 11 active sham with missing VADAS-cog values at 12, 18, and 24 weeks. These 18 subjects with all 3 primary time points missing discontinued the study. These values were multiply imputed from the longitudinal model as pre-specified.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Treatment Arm | Sham Arm
Number analyzed (Participants) | 95 | 95
score on a scale | -9.76 (1.54) | -5.31 (1.73)

2. Secondary Outcome: Number of Participants With Treatment Related Adverse Events as Assessed by MedDRA.
Time Frame: 24 weeks
Population: 3 participants from active sham group were migrated to treatment group.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm | Sham Arm
Number analyzed (Participants) | 98 | 92
Participants | 41 | 33

3. Secondary Outcome: Number of Participants With Treatment Related Serious Adverse Events as Assessed by MedDRA.
Time Frame: 24 weeks
Population: 3 participants from active sham group were migrated to treatment group.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm | Sham Arm
Number analyzed (Participants) | 98 | 92
Participants | 8 | 9

ADVERSE EVENTS:
Time Frame: The period from signing informed consent to the end of the study treatment follow-up (Month 12).
Description: 3 participants from active sham group were migrated to treatment group.
Arm/Group | Treatment Arm | Sham Arm
All-Cause Mortality (participants affected / at risk) | 0/98 | 1/92
Serious Adverse Events (participants affected / at risk) | 8/98 | 9/92
Other Adverse Events (participants affected / at risk) | 41/98 | 31/92
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm (N=98) | Sham Arm (N=92)
Endometrial Cancer (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest Pain (General disorders) | 1 (1) | 0 (0)
Coronavirus Infection (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (2) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Cervical Vertebral Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hip Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Amyotrophic Lateral Sclerosis (Nervous system disorders) | 1 (1) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Transient Ischemic Attack (Nervous system disorders) | 0 (0) | 1 (1)
Urinary Incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm (N=98) | Sham Arm (N=92)
Skin Irritation/Injury (Injury, poisoning and procedural complications) | 15 (20) | 3 (5)
Upper Respiratory Tract Infection (Infections and infestations) | 6 (7) | 7 (7)
Dehydration/Fluid Volume Decrease (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hypotension (Vascular disorders) | 0 (0) | 4 (4)
Diverticulitis (Infections and infestations) | 3 (3) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 5 (5) | 1 (1)
Gastrointestinal Upset (Gastrointestinal disorders) | 6 (6) | 0 (0)
Joint Pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Limb Fractures (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 6 (8) | 1 (1)
Nausea and Vomiting (Gastrointestinal disorders) | 3 (4) | 2 (3)
Dizziness (Nervous system disorders) | 3 (4) | 2 (2)
Non-Site Specific Injury (Injury, poisoning and procedural complications) | 3 (3) | 2 (5)
Supraventricular Arrhythmias (Cardiac disorders) | 3 (3) | 0 (0)
Dental pain (General disorders) | 0 (0) | 2 (2)
Headaches (Nervous system disorders) | 0 (0) | 2 (2)
Coughing (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Skin discomfort (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Infections, other (Infections and infestations) | 2 (2) | 0 (0)
Muscles/Tendon/Ligament injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Numbness/Tingling (Nervous system disorders) | 2 (2) | 0 (0)
Itch (Nervous system disorders) | 2 (2) | 0 (0)
Rate and Rhythm Disorders, Other (Cardiac disorders) | 2 (2) | 0 (0)
Site specific injuries, other (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Coronavirus Infection (Infections and infestations) | 2 (2) | 0 (0)
General pain and discomfort (General disorders) | 0 (0) | 2 (2)
Spinal Fractures (Injury, poisoning and procedural complications) | 0 (0) | 2 (4)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 2 (2)
Elevated Blood Pressure (Vascular disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2020-12-30): https://cdn.clinicaltrials.gov/large-docs/05/NCT03721705/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-03): https://cdn.clinicaltrials.gov/large-docs/05/NCT03721705/SAP_001.pdf
  • Informed Consent Form (2020-01-13): https://cdn.clinicaltrials.gov/large-docs/05/NCT03721705/ICF_002.pdf